CLINICAL TRIAL: NCT04405596
Title: Ambroxol as a Novel Disease Modifying Treatment for Lewy Body Dementia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Stephen Pasternak, Neurologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB:115252
Record Dates: First submitted 2020-04-29; First posted 2020-05-28 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lewy Body Disease
Keywords: Lewy Body Disease; Ambroxol; Cognition; Dementia
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — Ambroxol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambroxol (Experimental): Participants randomized to the 1350 mg/day group will begin with a dose of 450 mg, increasing bi-weekly to a dose of 1350 mg/day.
  Interventions: Drug: Ambroxol Hydrochloride
- Placebo (Placebo Comparator): Participants receive capsules visually identical to the experimental groups but without active ingredients.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ambroxol Hydrochloride — The treatment regimen consists of a titration phase and a maintenance phase. Participants begin the titration phase (Weeks 1 and 2) taking 6 capsules a day (450mg or 0 mg) divided BID (3 capsules in the morning and 3 capsules in the evening). The first medication dose will be taken at the end of Baseline visit and in the presence of the study Neurologist. Possible side effects will be observed for 30 minutes. Medication dose will increase bi-weekly to 12 capsules on Weeks 3 and 4, and 18 capsules on Weeks 5 and 6 divided BID. At the end of titration (Week 5) participants will have reached a maximum of 1350mg or 0mg per day, depending on group allocation. In the maintenance phase, participants will remain in their maximum dose (1350mg or 0mg) from Week 5 to Week 52 (End of Trial).
  Other Names: Mucosolvan
  Arms: Ambroxol
Other: Placebo — The treatment regimen consists of a titration phase and a maintenance phase. Participants begin the titration phase (Weeks 1 and 2) taking 6 capsules a day (450mg or 0 mg) divided BID (3 capsules in the morning and 3 capsules in the evening). The first medication dose will be taken at the end of Baseline visit and in the presence of the study Neurologist. Possible side effects will be observed for 30 minutes. Medication dose will increase bi-weekly to 12 capsules on Weeks 3 and 4, and 18 capsules on Weeks 5 and 6 divided BID. At the end of titration (Week 5) participants will have reached a maximum of 1350mg or 0mg per day, depending on group allocation. In the maintenance phase, participants will remain in their maximum dose (1350mg or 0mg) from Week 5 to Week 52 (End of Trial).
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind study investigating whether the medication Ambroxol is safe,effectiveness and well tolerated for the treatment of Lewy Body Dementia (LBD). Currently the main treatments for patients with LBD target symptom management. However, none of the medications treat the underlying cause of the disease, which includes the accumulation of protein in the brain. Therefore, even if patients respond well to symptomatic treatment, they continue to deteriorate. Therefore, the purpose of the current study is to make sure Ambroxol is safe to take long term and to test the effects of Ambroxol in treating the cognitive impairments associated with LBD by modifying the underlying causes of the disease.

There will be a total of 15 people participating this this study, which will last 52 weeks. Over the study period patients will undergo clinical, neuropsychological and neuroimaging assessment to assess changes.

DETAILED DESCRIPTION:
The increasing prevalence of dementia is a serious threat to our medical system and our society. About 500,000 Canadians are affected with dementia, and this number will rise to more than 1 million in the next 20 years. Dementia already costs our economy 15 billion dollars per year. While much of the focus of dementia is on Alzheimer's disease, autopsy studies suggest that up to 30% of dementia is due to diseases caused by abnormal alpha-synuclein accumulation (Synucleinopathies). In healthy brains, alpha-synuclein plays a number of important roles, especially in the process by which brain cells (neurons) communicate. However, when alpha-synuclein abnormally accumulates into clumps inside the neurons it forms Lewy bodies. Eventually, as a result, brain neurons will die causing widespread damage to specific brain regions.

Until the 1980's, cortical Lewy bodies were thought to be relatively rare. However, with improved alpha-synuclein immunostaining techniques, Lewy body dementias are now recognized as the second most common neurodegenerative dementia, after Alzheimer's disease. Lewy body-related disorders include idiopathic Parkinson's disease (PD), Parkinson's disease dementia (PDD) and Lewy Body Dementia (LBD). In LBD, alpha- synuclein accumulation is found in the brainstem, limbic and neocortical regions, giving rise to autonomic, cognitive and motor impairments.

Cognitive Symptoms: Progressive cognitive decline typically begins early in the course of the disease in advance of parkinsonism, but by consensus may follow the development of motor signs up to 1 year. Impaired cognitive domains include executive and visual-spatial functions, attention and short-term memory. For example, patients may have difficulty multi-tasking, following conversations, episodes of staring and perturbed flow of ideas. Regarding short-term memory, patients with LBD experience impairment in memory retrieval, which can be improved by cueing, which is in contrast to memory encoding seen in AD. The early presence of recurrent visual hallucinations is also common in patients with LBD and therefore diagnostically useful. Later in the course of the disease, delusions can be present giving rise to paranoia.

Motor symptoms: Parkinsonian motor signs in LBD are often symmetric, with bradykinesia and gait impairments being more common than resting tremor. Importantly, patients with LBD will often show limited or no response to typical Parkinson's disease pharmacological intervention such as levodopa/carbidopa. LBD patients however do show reduced dopamine transporter activity on single-photon emission computed tomography (SPECT) or positron emission tomography (PET) imaging.

Other Associated symptoms can include: loss of olfaction, autonomic dysfunction (i.e. neurogenic orthostatic hypotension, constipation, neurogenic urinary frequency and urgency), high sensitivity to medications and rapid eye movement sleep behaviour disorder typically reported by a sleep partner as kicking, punching, yelling and acting out their dreams.

Mechanism for targeting Lewy bodies: A potential target for disease-modifying treatment is the enzyme β-Glucocerebrosidase (GCase; gene name GBA1). Glucocerebrosidase (GCase) is a degradative enzyme that resides in a subcellular compartment called the lysosome, and cleaves a neutral glycolipid, glucocerebroside, present in the plasma membrane of most cells. GCase is intimately linked with Parkinson's disease - a Lewy body-related disorder. Being an "asymptomatic carrier" of a GCase mutation is currently the highest genetic risk factor for Parkinson's disease, Parkinson's disease dementia and Lewy Body Dementia, with some studies suggesting up to 1/3 of patients carry mutations. Reductions in GCase activity most likely also play a role in sporadic Parkinson's disease, as these patients have lower levels of GCase in their brain and cerebrospinal fluid, even when they do not carry a mutant GCase allele. Laboratory studies have demonstrated a direct link between GCase activity and α-synuclein accumulation. In cultured cells, loss of GCase results in α-synuclein accumulation and this process feeds back upon itself, with overexpression of α-synuclein further inhibiting GCase function, and increasing GCase expression reducing α-synuclein. Moreover, reducing GCase genetically or pharmacologically in animal studies results in increased α-synuclein aggregates. Remarkably, overexpressing GCase in the brain of a Parkinson's disease mouse model reduces α-synuclein and improves cognition. Taken together, these findings suggest that increasing GCase levels could be a therapy that addresses the underlying pathophysiology of Lewy body-related disorders such as Lewy Body dementia to modify the course of disease progression.

Background on Ambroxol Studies: Ambroxol is an expectorant that has been available over the counter in more than 50 countries for over 30 years. The Mahuran Lab identified Ambroxol by screening a library of compounds as an agent that stabilizes wild-type (normal) GCase. By stabilizing GCase, Ambroxol is able to markedly increase GCase protein and activity in normal and Gaucher disease fibroblasts at doses of 10 µM. Ambroxol can also increase GCase in normal mouse neuronal cultures to more than 150% of normal at a dose of 30 µM. Ambroxol has good lipophilicity (cLogP = 2.8) and low polar surface area (PSA 58 Å2), predicting good CNS penetration. Unpublished studies performed by ExSAR corporation demonstrate that in single and multiple dose experiments in rats, Ambroxol crossed rapidly into the brain and exhibited brain to plasma concentration ratios of greater than 10 indicating outstanding CNS penetration. In pilot studies, Ambroxol was effective at improving GCase function in humans. In a trial aimed at non-neurological Gaucher disease, 12 patients received 150 mg/day for 6 months, and all but one had some measurable improvement. The best response was in the lightest patient (who received 3 mg/kg/day), suggesting that Ambroxol was under dosed. Ambroxol has also been administered to three Japanese Gaucher disease patients with severe neurological disease, at 1000-3000 mg/day for 12-31 months. These patients had improvements in seizure frequency and neurological symptoms; one patient regained the ability to sit unsupported and to walk. Importantly, in a recent study of Ambroxol in 18 Parkinson's disease patients, the authors observed a 35% increase in CSF GCase protein levels at a daily dose of 1260mg with no serious adverse events.

Safety: Ambroxol has an excellent safety record, and has been studied in >15,000 patients in more than 100 trials. Ambroxol is sold over the counter in much of the world as an expectorant at doses of 75-120 mg/day. Ambroxol is considered so safe that it is approved for intravenous use in pregnant women at a dose of 1000 mg/day IV (15 mg/kg) to improve fetal lung maturation before preterm delivery. Clinical trials in more than 390 pregnant women have been performed using doses up to 3000 mg in one day and 1300 mg/day for up to 33 days. Critically ill neonates have also been given doses as high as 30 mg/kg for respiratory distress. The fact that Ambroxol has been used at very high doses in pregnant women and neonates suggests that these doses are safe.

Project Summary: This is a proof of principle randomized, placebo-controlled, double-blind study investigating whether the medication Ambroxol (dose: 1350mg/day) is safe, well tolerated and will raise GCase levels in the CSF and plasma of patients diagnosed with probable Lewy Body Dementia (LBD). Additionally, increased levels of the enzyme β-glucocerebrosidase (GCase) and lower the levels of the protein α-synuclein have both been shown to improve cognition in mouse models. Therefore, as secondary aim will be to investigate whether Ambroxol will improve cognitive symptoms in patients diagnosed with Lewy Body Dementia (LBD). This will be a 52-week trial of Ambroxol in 15 patients diagnosed with probable LBD. Patients will undergo clinical, neuropsychological and neuroimaging assessment throughout the study to assess changes. Ambroxol has never been examined in LBD patients; however, trials of pharmacological chaperone therapy have been suggested in a recent review in the journal "The Proceedings of the National Academy of Sciences". A successful outcome of this trial will greatly accelerate the development of therapeutics for neurodegenerative disease. This proposal outlines a completely novel pharmacological target for LBD, namely the GCase enzyme. The investigators also propose a completely novel therapy using the drug Ambroxol, an agent considered safe enough to give to pregnant women, which has improved GCase function in pilot studies in humans. This strategy could stabilize the underlying pathology of Lewy Body Dementia; it might allow patients to get better. Furthermore, repurposing an existing medication with excellent safety record will greatly shorten the time to bring this therapy to general use, allowing us to leapfrog the normally decades-long drug development process.

ELIGIBILITY:
Inclusion Criteria:

1. Probable diagnosis of Lewy Body Dementia
2. Age greater than 50 years old
3. Montreal Cognitive Assessment (MoCA) score: 24-18
4. Patients must have a responsible caregiver = 4days/week
5. Must be on a stable dose of medications for parkinsonism (levodopa, dopaminergic agonist) and cognition (cholinesterase inhibitors) and psychiatric (i.e. antidepressants, antipsychotic) for at least 3 months prior to the study

Exclusion Criteria:

1. Evidence of stroke or other neurological condition
2. Any other serious underlying condition or brain disorder that can account in part of in full for the clinical presentation (i.e. cancer or unstable cardiac disease etc.)
3. Contraindication to MRI e.g. presence of metal fragments in head or eye, implanted electrical devices or conductive implants or devices (pacemakers, neurostimulators).
4. Unable to undergo DAT-scan
5. Depression that is, in the opinion of the investigator, significant enough to interfere with neuropsychology and safety assessments
6. Females who are pregnant or breastfeeding, or planning to conceive within the study period
7. Concurrent treatment with oral anticoagulants (including Vitamin K agonists and Novel Oral Anticoagulants (NOACs)) within 4 weeks of screening or anticipated during the 52 week double-blind and open label periods. Specifically, Apixaban, Dabigatran, Edoxaban, Fondaparinux, Rivaroxaban, and Warfarin are prohibited concomitant medications. Exceptions: antiplatelet agents such as Aspirin, Clopidogrel, and Aggrenox.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mini Mental State Examination score from baseline over time | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Monitor safety using frequent cognitive evaluations using the mini mental state examination. Lower scores are indicative of worsening cognitive impairment [score range: 0-30]
Change in the incidence, nature and severity of AE's and SAE's from baseline | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Change in the number of participants with AE's and SAE's
Change in the number of participants with treatment discontinuations and study discontinuation due to AEs from baseline | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Change from baseline in the number of participants with treatment and/or study discontinuation will be used to demonstrate safety and tolerability
Change in the number of participants with electrocardiogram (ECG) abnormalities | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Change from baseline in the number of participants with clinically significant ECG abnormalities (QT interval) to demonstrate safety
Change from baseline the number of participants with abnormal changes in hemodynamic values while seated | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Changes in hemodynamic values from baseline over time to demonstrate safety
Change from baseline the number of participants with abnormal changes in hemodynamic values while standing | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Changes in hemodynamic values from baseline over time to demonstrate safety
Change in blood analyses from baseline over time | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Change from baseline in number of participants with abnormal changes in clinical laboratory blood tests from baseline over time for safety
Change in urine analyses from baseline over time | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Change from baseline in number of participants with abnormal changes in clinical laboratory urine tests from baseline over time for safety
Change from baseline in plasma concentrations of Ambroxol from blood sample | Baseline, week 4, week 10, week 26, week 52
  Change in plasma Ambroxol concentrations from blood sample from baseline
Change from baseline in cerebrospinal fluid (CSF) concentrations of Ambroxol at specified time points | Baseline, week 10, week 52
  Change in Ambroxol concentrations from cerebrospinal fluid sample from baseline
Change from baseline in enzyme β-Glucocerebrosidase (GCase) concentration levels in CSF | Baseline, week 10, week 52
  Change in GCase concentration in the CSF from baseline
Change from baseline in enzyme β-Glucocerebrosidase (GCase) concentration levels in white blood cells | Baseline, week 4, week 10, week 26, week 52
  Change in white blood cell GCase concentrations from baseline

SECONDARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline, week 26, and week 52
  Demonstrate the efficacy of Ambroxol in improving, or slowing the progression of cognitive deficits. Lower scores are indicative of worsening cognitive function [score range: 40-160]
Clinician's Global Impression of Change (CGIC) | Baseline, week 26, and week 52
  Demonstrate the efficacy of Ambroxol in improving, or slowing the progression of cognitive deficits. Patients are assessed as: no change, minimal, moderate and marked worsening, minimal, moderate and marked improvement
Montreal Cognitive Assessment (MoCA) | Baseline, week 26, and week 52
  Demonstrate the efficacy of Ambroxol in improving, or slowing the progression of cognitive deficits. Lower scores are indicative of worsening cognitive impairment [score range: 0-30]
Trail making test A and B to assess cognitive function | Baseline, week 26, and week 52
  Demonstrate the efficacy of Ambroxol in improving, or slowing the progression of cognitive deficits: Higher times to complete are indicative of worsening cognitive function [Max time: 300 seconds]
Parkinson's disease - Cognitive rating scale to assess cognitive function | Baseline, week 26, and week 52
  Demonstrate the efficacy of Ambroxol in improving, or slowing the progression of cognitive deficits. Lower scores are indicative of higher cognitive dysfunction [Score range: 0-134]
Change in regional brain magnetic resonance imaging atrophy measures | Baseline, week 52
  Change in hippocampal atrophy (cm3)
Change in global brain magnetic resonance imaging atrophy measures | Baseline, week 52
  Change in brain ventricle volume (cm3)
Change in plasma biomarkers | Baseline, week 4, week 10, week 18, week 26, week 34, week 42, week 52
  Change in levels of plasma biomarkers: α-synuclein (pg/ml), Tau (pg/ml), phospho-Tau (pg/ml) and beta amyloid-42 (pg/ml) in plasma
Change in Cerebrospinal Fluid (CSF) biomarkers | Baseline, week 10, week 52
  Change in levels of CSF biomarkers: α-synuclein (pg/ml), Tau (pg/ml), phospho-Tau (pg/ml) and beta amyloid-42 (pg/ml) in CSF
Neuropsychological Inventory (NPI) | Baseline, week 26, and week 52
  Demonstrate change or slowed progression in standard tests of mood and neuropsychiatric symptoms. Assesses frequency and severity of neuropsychological symptoms with higher scores indicative of more symptoms, higher frequency and more severe. [Score range: 0-144]
Geriatric Depression Scale | Baseline, week 26, and week 52
  Demonstrate change or slowed progression in standard tests of mood and neuropsychiatric symptoms: Higher scores indicate more severe depression [score range: 0-15]
The Motor subscale of Unified Parkinson's Disease Rating Scale (UPDRS-III) | Baseline, week 26, and week 52
  Demonstrate change or slowed progression in tests of motor function/Parkinsonism: Higher scores indicate more dysfunction [score range: 0-108]
Timed Up and Go | Baseline, week 26, and week 52
  Demonstrate change or slowed progression in tests of motor function/Parkinsonism. Higher times indicate slower movement and more motor impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Parkwood Institute, London, Ontario, Canada

REFERENCES:
- [Background] Bendor JT, Logan TP, Edwards RH. The function of alpha-synuclein. Neuron. 2013 Sep 18;79(6):1044-66. doi: 10.1016/j.neuron.2013.09.004. PMID 24050397
- [Background] Gomperts SN. Lewy Body Dementias: Dementia With Lewy Bodies and Parkinson Disease Dementia. Continuum (Minneap Minn). 2016 Apr;22(2 Dementia):435-63. doi: 10.1212/CON.0000000000000309. PMID 27042903
- [Background] Balducci C, Pierguidi L, Persichetti E, Parnetti L, Sbaragli M, Tassi C, Orlacchio A, Calabresi P, Beccari T, Rossi A. Lysosomal hydrolases in cerebrospinal fluid from subjects with Parkinson's disease. Mov Disord. 2007 Jul 30;22(10):1481-1484. doi: 10.1002/mds.21399. PMID 17546678
- [Background] Gegg ME, Burke D, Heales SJ, Cooper JM, Hardy J, Wood NW, Schapira AH. Glucocerebrosidase deficiency in substantia nigra of parkinson disease brains. Ann Neurol. 2012 Sep;72(3):455-63. doi: 10.1002/ana.23614. PMID 23034917
- [Background] Laoag-Fernandez JB, Fernandez AM, Maruo T. Antenatal use of ambroxol for the prevention of infant respiratory distress syndrome. J Obstet Gynaecol Res. 2000 Aug;26(4):307-12. doi: 10.1111/j.1447-0756.2000.tb01327.x. PMID 11049243
- [Background] Luan Z, Li L, Higaki K, Nanba E, Suzuki Y, Ohno K. The chaperone activity and toxicity of ambroxol on Gaucher cells and normal mice. Brain Dev. 2013 Apr;35(4):317-22. doi: 10.1016/j.braindev.2012.05.008. Epub 2012 Jun 7. PMID 22682976
- [Background] Luerti M, Lazzarin A, Corbella E, Zavattini G. An alternative to steroids for prevention of respiratory distress syndrome (RDS): multicenter controlled study to compare ambroxol and betamethasone. J Perinat Med. 1987;15(3):227-38. doi: 10.1515/jpme.1987.15.3.227. PMID 3323457
- [Background] Maegawa GH, Tropak MB, Buttner JD, Rigat BA, Fuller M, Pandit D, Tang L, Kornhaber GJ, Hamuro Y, Clarke JT, Mahuran DJ. Identification and characterization of ambroxol as an enzyme enhancement agent for Gaucher disease. J Biol Chem. 2009 Aug 28;284(35):23502-16. doi: 10.1074/jbc.M109.012393. Epub 2009 Jul 3. PMID 19578116
- [Background] Malerba M, Ragnoli B. Ambroxol in the 21st century: pharmacological and clinical update. Expert Opin Drug Metab Toxicol. 2008 Aug;4(8):1119-29. doi: 10.1517/17425255.4.8.1119. PMID 18680446
- [Background] Manning-Bog AB, Schule B, Langston JW. Alpha-synuclein-glucocerebrosidase interactions in pharmacological Gaucher models: a biological link between Gaucher disease and parkinsonism. Neurotoxicology. 2009 Nov;30(6):1127-32. doi: 10.1016/j.neuro.2009.06.009. Epub 2009 Jul 2. PMID 19576930
- [Background] Mazzulli JR, Xu YH, Sun Y, Knight AL, McLean PJ, Caldwell GA, Sidransky E, Grabowski GA, Krainc D. Gaucher disease glucocerebrosidase and alpha-synuclein form a bidirectional pathogenic loop in synucleinopathies. Cell. 2011 Jul 8;146(1):37-52. doi: 10.1016/j.cell.2011.06.001. Epub 2011 Jun 23. PMID 21700325
- [Background] Mullin S, Smith L, Lee K, D'Souza G, Woodgate P, Elflein J, Hallqvist J, Toffoli M, Streeter A, Hosking J, Heywood WE, Khengar R, Campbell P, Hehir J, Cable S, Mills K, Zetterberg H, Limousin P, Libri V, Foltynie T, Schapira AHV. Ambroxol for the Treatment of Patients With Parkinson Disease With and Without Glucocerebrosidase Gene Mutations: A Nonrandomized, Noncontrolled Trial. JAMA Neurol. 2020 Apr 1;77(4):427-434. doi: 10.1001/jamaneurol.2019.4611. PMID 31930374
- [Background] Nalls MA, Duran R, Lopez G, Kurzawa-Akanbi M, McKeith IG, Chinnery PF, Morris CM, Theuns J, Crosiers D, Cras P, Engelborghs S, De Deyn PP, Van Broeckhoven C, Mann DM, Snowden J, Pickering-Brown S, Halliwell N, Davidson Y, Gibbons L, Harris J, Sheerin UM, Bras J, Hardy J, Clark L, Marder K, Honig LS, Berg D, Maetzler W, Brockmann K, Gasser T, Novellino F, Quattrone A, Annesi G, De Marco EV, Rogaeva E, Masellis M, Black SE, Bilbao JM, Foroud T, Ghetti B, Nichols WC, Pankratz N, Halliday G, Lesage S, Klebe S, Durr A, Duyckaerts C, Brice A, Giasson BI, Trojanowski JQ, Hurtig HI, Tayebi N, Landazabal C, Knight MA, Keller M, Singleton AB, Wolfsberg TG, Sidransky E. A multicenter study of glucocerebrosidase mutations in dementia with Lewy bodies. JAMA Neurol. 2013 Jun;70(6):727-35. doi: 10.1001/jamaneurol.2013.1925. PMID 23588557
- [Background] Narita A, Shirai K, Itamura S, Matsuda A, Ishihara A, Matsushita K, Fukuda C, Kubota N, Takayama R, Shigematsu H, Hayashi A, Kumada T, Yuge K, Watanabe Y, Kosugi S, Nishida H, Kimura Y, Endo Y, Higaki K, Nanba E, Nishimura Y, Tamasaki A, Togawa M, Saito Y, Maegaki Y, Ohno K, Suzuki Y. Ambroxol chaperone therapy for neuronopathic Gaucher disease: A pilot study. Ann Clin Transl Neurol. 2016 Feb 2;3(3):200-15. doi: 10.1002/acn3.292. eCollection 2016 Mar. PMID 27042680
- [Background] Sardi SP, Clarke J, Kinnecom C, Tamsett TJ, Li L, Stanek LM, Passini MA, Grabowski GA, Schlossmacher MG, Sidman RL, Cheng SH, Shihabuddin LS. CNS expression of glucocerebrosidase corrects alpha-synuclein pathology and memory in a mouse model of Gaucher-related synucleinopathy. Proc Natl Acad Sci U S A. 2011 Jul 19;108(29):12101-6. doi: 10.1073/pnas.1108197108. Epub 2011 Jul 5. PMID 21730160
- [Background] Sardi SP, Clarke J, Viel C, Chan M, Tamsett TJ, Treleaven CM, Bu J, Sweet L, Passini MA, Dodge JC, Yu WH, Sidman RL, Cheng SH, Shihabuddin LS. Augmenting CNS glucocerebrosidase activity as a therapeutic strategy for parkinsonism and other Gaucher-related synucleinopathies. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):3537-42. doi: 10.1073/pnas.1220464110. Epub 2013 Jan 7. PMID 23297226
- [Background] Schapira AH, Gegg ME. Glucocerebrosidase in the pathogenesis and treatment of Parkinson disease. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):3214-5. doi: 10.1073/pnas.1300822110. Epub 2013 Feb 14. No abstract available. PMID 23412333
- [Background] Schmalisch G, Wauer RR, Bohme B. Changes in pulmonary function in preterm infants recovering from RDS following early treatment with ambroxol: results of a randomized trial. Pediatr Pulmonol. 1999 Feb;27(2):104-12. doi: 10.1002/(sici)1099-0496(199902)27:23.0.co;2-t. PMID 10088933
- [Background] Wauer RR, Schmalisch G, Hammer H, Buttenberg S, Weigel H, Huth M. Ambroxol for prevention and treatment of hyaline membrane disease. Eur Respir J Suppl. 1989 Mar;3:57S-65S. PMID 2662997
- [Background] Zimran A, Altarescu G, Elstein D. Pilot study using ambroxol as a pharmacological chaperone in type 1 Gaucher disease. Blood Cells Mol Dis. 2013 Feb;50(2):134-7. doi: 10.1016/j.bcmd.2012.09.006. Epub 2012 Oct 22. PMID 23085429
- [Background] Low, P., & Benarroch, E. (2008). Clinical Autonomic Disorders. (P. Low & E. Benarroch, Eds.) (Third). Philadelphia: Wolters Kluwer Health/Lippincott Williams & Wilkins
- [Background] Narita, A., Zhou, L., Higaki, K., Togawa, M., Maegaki, Y., Nanba, E., … Ohno, K. (2012). Chemical chaperone therapy for neuropathic Gaucher disease. In 12th International Child Neurology Congress and the 11th Asian and Oceanian Congress of Child Neurology Brisbane (pp. 50-5)